CLINICAL TRIAL: NCT06784999
Title: Randomized Prospective Study Comparing Sufentanil Infusion vs Intravenous Methadone for Postoperative Analgesia Following Head and Neck Dissection With Free Flap or Rotational Reconstruction
Brief Title: Sufentanil Infusion vs Intravenous Methadone for Postoperative Analgesia Following Head and Neck Dissection With Free Flap or Rotational Reconstruction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Gulraj Chawla, MD, Assistant Professor of Clinical Anesthesia Program Director, Regional Anesthesia and Acute Pain Medicine Fellowship, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21583
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Free Flap Reconstruction
Keywords: head and neck dissection; free flap; sufentanil; methadone
MeSH Terms: interventions — Sufentanil; Methadone

STUDY DESIGN:
Intervention Model Description: A total of 128 subjects will be randomized by a computer program into two groups.
  1. Intravenous Sufentanil - 0.5 mcg /kg/min ideal body weight N=64
  2. Intravenous Methadone - 0.2 mcg/kg ideal body weight max dose of 20mg N=64
Who Masked: Participant, Outcomes Assessor
Masking Description: The Primary investigator or his/her designee will inform the anesthesiology team caring for each subject of the am of the study they are in for each case. Subjects and research staff doing post operative assessments will be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sufentanil (Other): 1. Intravenous sufentanil starting at a dose of 0.5 mcg/kg/min hr ideal body weight (IBW) at the beginning of the case, prior to surgical incision, with a discontinuation of the infusion when the surgical microscope is removed from the patient field and the closure of the incision(s) begins. (n=64)
  Interventions: Drug: sufentanil
- Methadone (Other): 2. Intravenous methadone of 0.2 mg/kg IBW up to a maximum dose of 20mg, rounded to the nearest milligram. The methadone will be given at the beginning of the case, prior to surgical incision. n=64)
  Interventions: Drug: methadone

INTERVENTIONS:
Drug: sufentanil — 1. Intravenous sufentanil starting at a dose of 0.5 mcg/kg/min hr ideal body weight (IBW) at the beginning of the case, prior to surgical incision, with a discontinuation of the infusion when the surgical microscope is removed from the patient field and the closure of the incision(s) begins. (n=64)
  Arms: Sufentanil
Drug: methadone — 2. Intravenous methadone of 0.2 mg/kg IBW up to a maximum dose of 20mg, rounded to the nearest milligram. The methadone will be given at the beginning of the case, prior to surgical incision. n=64)
  Arms: Methadone

SUMMARY:
The main purpose of this study is to determine which type of medication, sufentanil or methadone, is better at controlling pain during and, more importantly, after surgery in patients undergoing a head and neck dissection with free flap or rotational tissue reconstruction. Prior to their operation, subjects will be randomized to receive either Sufentanil or Methadone. After surgery, research staff will obtain information about recovery and pain levels.

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing head and neck dissection with free flap or rotational reconstruction at Indiana University Health Adult Academic Health Center

  * ASA class 1, 2, or 3 (See Appendix)
  * Age 18 to 80
  * male or female
  * Able and willing to provide written informed consent

Exclusion Criteria:

* Any contraindication to opiates, (i.e. allergy to opioids, substance use disorder) as determined by PI review and any contraindications reported by the patient
* Patient on home methadone at any dose
* Any physical, mental or medical conditions which, in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery
* Known true allergy to the study medications (sufentanil, methadone)
* Any history of substance abuse in the past 6 months which would include heroin or any other illegal street drugs
* End stage liver disease, end stage renal disease
* Patient staying intubated or on mechanical ventilation after surgery
* Patient (home dose) taking more than 30mg PO morphine equivalent (OME) per day
* Any additional and concurrent surgical procedures to the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
IV morphine equivalent | 24 hours
  Cumulative milligrams IV morphine equivalent

SECONDARY OUTCOMES:
Opioid Consumption | 1 hour after arrival time in post anesthesia care unit
  Opioid Consumption and morphine equivalent (MME)
Opioid Consumption | 12 hour after arrival time in post anesthesia care unit
  Opioid Consumption and morphine equivalent (MME)
Opioid Consumption | 24 hour after arrival time in post anesthesia care unit
  Opioid Consumption and morphine equivalent (MME)
Pain Scores | 1 hour after arrival time in post anesthesia care unit
  Visual analog scale (VAS) pain score on a scale of 1-10 (increments of 1 unit), 1 being no pain at all and 10 being the most pain the patient has ever experienced
Pain Scores | 12 hour after arrival time in post anesthesia care unit
  Visual analog scale (VAS) pain score on a scale of 1-10 (increments of 1 unit), 1 being no pain at all and 10 being the most pain the patient has ever experienced
Pain Scores | 24 hour after arrival time in post anesthesia care unit
  Visual analog scale (VAS) pain score on a scale of 1-10 (increments of 1 unit), 1 being no pain at all and 10 being the most pain the patient has ever experienced
Opioid side effect - Nausea | After arrival time to post anesthesia care unit until 24 hrs./completion of study
  Incident of opioid side effect - Nausea
Opioid side effect - Puritis | After arrival time to post anesthesia care unit until 24 hrs./completion of study
  Incident of opioid side effect - Puritis
Opioid side effect - Respiratory Depression | After arrival time to post anesthesia care unit until 24 hrs./completion of study
  Incident of opioid side effect - Respiratory Depression

CONTACTS AND LOCATIONS:
Overall Officials: Gulraj S Chawla, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No